CLINICAL TRIAL: NCT07358143
Title: Associations Between Motor Ability and Adaptive Behavior and Their Predictive Value in Children With Severe Intellectual Disability
Brief Title: Gross Motor Skills Predict Adaptive Behavior in Institutionalized Children With Severe Intellectual Disability: A Cross-Sectional Study
Acronym: TGMD-ADQ
Status: Completed | Type: Observational
Sponsor: Xili Wen (Other)
Responsible Party: Sponsor-Investigator, Xili Wen, Ph.DStudent, Shanghai University of Sport
Organization: Shanghai University of Sport (Other)
Other Study IDs: 102772024RT062; SUS (Other: Shanghai University of Sport)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Severe Intellectual Disability
Keywords: Intellectual Disability; Adaptive Behavior; Gross Motor Skills; Motor Competence
MeSH Terms: conditions — Intellectual Disability | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe ID Cohort (Institutionalized Children): A convenience sample of 227 orphaned children with severe intellectual disability recruited from six social welfare institutions (orphanages) in China. All participants resided in institutional care for extended periods and completed one-time assessments, including TGMD-2 motor testing and caregiver-assisted ADQ adaptive behavior evaluation. Data were collected between May and June 2024.
  Interventions: Diagnostic Test: Test of Gross Motor Development-Second Edition (TGMD-2) Assessment; Diagnostic Test: Adaptive Behavior Questionnaire for Children (ADQ) Assessment

INTERVENTIONS:
Diagnostic Test: Test of Gross Motor Development-Second Edition (TGMD-2) Assessment — Standardized gross motor skill assessment (locomotor and object control subtests) administered at a single time point. Testing followed an instruction-demonstration-imitation protocol; sessions were video recorded and independently scored by two trained raters with adjudication by a third rater if needed. This is an assessment procedure, not a therapeutic intervention.
Diagnostic Test: Adaptive Behavior Questionnaire for Children (ADQ) Assessment — Caregiver-assisted administration of the Adaptive Behavior Questionnaire for Children (ADQ) to obtain the overall ADQ Index and domain scores (independence, cognition, socialization). Standardized scoring was used; ADQ Index < 70 was used to classify low adaptive behavior for analysis. This is an assessment procedure, not a therapeutic intervention.

SUMMARY:
This study examines whether gross motor skills are linked to everyday functioning (adaptive behavior) in children with severe intellectual disability (ID) living in social welfare institutions. We recruited 227 orphaned children aged 6-12 years from six welfare institutions in China.

Gross motor competence was assessed using the Test of Gross Motor Development-Second Edition (TGMD-2), which includes locomotor skills and object control skills. :contentReference[oaicite:1]{index=1} Adaptive behavior was assessed using the Adaptive Behavior Questionnaire for Children (ADQ), which provides an overall ADQ Index and scores for independence, cognition, and socialization.

Assessments were conducted on site by a trained research team between May and June 2024. TGMD-2 sessions were video recorded and scored by trained raters, and caregivers completed the ADQ with assistance to ensure completeness. :contentReference[oaicite:3]{index=3} We will evaluate associations between TGMD-2 scores and ADQ outcomes and assess whether the TGMD-2 total score can help screen for children at risk of low adaptive functioning (ADQ Index < 70).

All procedures were approved by the local university ethics committee (approval number: 102772024RT062), and informed consent was obtained from institutional administrators and caregivers.

DETAILED DESCRIPTION:
Background:

Children with severe intellectual disability (ID) living in institutional settings often experience substantial limitations in both motor competence and adaptive functioning. Efficient ways to identify children at higher functional risk may help guide prioritization of supportive services within resource-limited institutions.

Study Design:

This is an observational, cross-sectional study conducted in six social welfare institutions (orphanages) in China using a convenience sampling approach. A total of 227 orphaned children aged 6-12 years with severe ID were recruited. Severe ID was defined based on DSM-5 clinical diagnosis with standardized intelligence test scores ranging from 20 to 34. Additional inclusion criteria included basic auditory and visual abilities and the capacity to follow simple motor instructions. Exclusion criteria included severe musculoskeletal disorders, neurological comorbidities (e.g., active epilepsy), other physical conditions limiting motor assessment participation, or major surgery within the previous six months.

Procedures and Assessments:

All assessments were conducted on site by a professionally trained research team between May and June 2024. :contentReference[oaicite:9]{index=9} Gross motor competence was measured using the Test of Gross Motor Development-Second Edition (TGMD-2), which includes locomotor and object control subtests. Testing followed a standardized instruction-demonstration-imitation protocol. TGMD-2 sessions were video recorded; two trained raters independently scored performance, and a third rater adjudicated disagreements to enhance scoring accuracy.

Adaptive behavior was assessed using the Adaptive Behavior Questionnaire for Children (ADQ), which includes three domains (independence, cognition, and socialization) and yields an overall Adaptive Deviation Quotient (ADQ Index) based on standardized scoring procedures. An ADQ Index < 70 was used to classify low adaptive behavior. The ADQ was completed with face-to-face assistance provided to caregivers to ensure data completeness and reliability.

Analysis Plan:

Descriptive statistics will summarize participant characteristics. Pearson correlations will examine associations between TGMD-2 scores (total and subtests) and ADQ outcomes. Multiple linear regression models will evaluate the unique contribution of TGMD-2 scores to overall adaptive functioning and ADQ domains while adjusting for age and sex. Receiver operating characteristic (ROC) analysis will be used to evaluate the ability of TGMD-2 total score to identify low adaptive behavior (ADQ Index < 70) and to estimate an optimal screening threshold using standard ROC indices.

Ethics:

All procedures were conducted in accordance with the Declaration of Helsinki and approved by the local university ethics committee (approval number: 102772024RT062). Written informed consent was obtained from institutional administrators and caregivers.

ELIGIBILITY:
Inclusion Criteria:1.Clinical diagnosis of severe intellectual disability according to DSM-5, with standardized intelligence test scores ranging from 20 to 34.2.Age between 6 and 12 years.3.Basic auditory and visual abilities and the capacity to understand and follow simple motor instructions.4.Orphaned children residing in social welfare institutions (orphanages) for extended periods.5.Written informed consent obtained from institutional administrators and caregivers.

Exclusion Criteria:1.Severe musculoskeletal disorders, neurological comorbidities (e.g., active epilepsy), or other physical conditions that could restrict participation in gross motor assessments.2.History of major surgery within the previous six months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A convenience sample of 227 orphaned children with severe intellectual disability (DSM-5; IQ 20-34), aged 6-12 years, recruited from six social welfare institutions (orphanages) in China. All participants resided in institutional care for extended periods and completed one-time on-site assessments, including TGMD-2 gross motor testing and caregiver-assisted ADQ adaptive behavior evaluation. Data were collected between May and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Adaptive behavior (ADQ Index) | At assessment (single time point; May-June 2024).
  Overall adaptive functioning measured by the Adaptive Behavior Questionnaire for Children (ADQ). The ADQ Index is derived from standardized scoring procedures; higher scores indicate better adaptive behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Sport, School of Physical Education and Training, Shanghai, Ph.d, China

IPD SHARING:
Plan to Share IPD: No